CLINICAL TRIAL: NCT02738450
Title: A Phase Ib Multi-Center, Double-Blind, Randomized, Placebo-Controlled Dose Escalation Study of the Safety, Tolerability and Immunogenicity of ACI-24 in Adults With Down Syndrome
Brief Title: Safety, Tolerability and Immunogenicity of ACI-24 Vaccine in Adults With Down Syndrome
Acronym: 3-Star
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Disease Cooperative Study (ADCS) (Other); LuMind IDSC Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACI-24-1301; 1R01AG047922-01 (NIH)
Record Dates: First submitted 2016-04-01; First posted 2016-04-14 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Down Syndrome
Keywords: cognitive decline
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACI-24 low dose (Active Comparator): Vaccine formulation will be administrated s.c. 7 times.
  Interventions: Biological: ACI-24 low dose
- ACI-24 high dose (Active Comparator): Vaccine formulation will be administrated s.c. 7 times.
  Interventions: Biological: ACI-24 high dose
- Placebo (Placebo Comparator): The placebo is ready-to-use solution for injection, administrated s.c. 7 times.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACI-24 low dose — ACI-24 administered as a sterile suspension in PBS via s.c. injection.
  Arms: ACI-24 low dose
Biological: ACI-24 high dose — ACI-24 administered as a sterile suspension in PBS via s.c. injection.
  Arms: ACI-24 high dose
Biological: Placebo — Placebo is a standard PBS sterile solution administrated via s.c. injection.
  Other Names: PBS
  Arms: Placebo

SUMMARY:
The purpose of this study is to test in adults with Down Syndrome the safety, tolerability and immunogenicity of a vaccine, ACI-24.

DETAILED DESCRIPTION:
This is a prospective multi-center, placebo controlled, double-blind and randomized dose escalation study of 2 doses of ACI-24 versus Placebo over 24 months with a total of 21 visits.

All subjects will receive the study medication (ACI-24 or Placebo) 7 times via s.c. injection (12 months) and will be followed up for 12 months after the last dose with a final safety and efficacy assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with Down Syndrome aged ≥25 to ≤45 years, with a cytogenetic diagnosis being either Trisomy 21 or Complete Unbalanced Translocation of the Chromosome 21.
* Subjects and their study partner/legal representative in the opinion of the investigator able to understand and to provide written informed consent.
* Written informed consent obtained from subjects and their study partner/legal representative before any trial-related activities.
* In the opinion of the investigator able to fully participate in the trial and sufficiently proficient in English to be capable of reliably completing study assessments.
* Subjects have a study partner/legal representative who have direct contact with the subjects at least 10 hours per week and who can be asked questions about the subjects.

Exclusion Criteria:

* Subjects weighing less than 40 kg.
* IQ less than 40 (as assessed by Kaufman Brief Intelligence Test, Second Edition (KBIT-2).
* In the investigators opinion, any clinically significant current psychiatric or neurologic illness, including a past illness with a risk of recurrence, other than Down syndrome.
* Any medical condition likely to significantly hamper the evaluation of safety of the study drug.
* DSM-IV criteria for drug or alcohol abuse or dependence currently met within the past five years.
* History or presence of uncontrolled seizures. If history of seizures, they must be well controlled with no occurrence of seizures in the past 2 years prior to study screening. The use of anti-epileptic medications is permitted.
* History of meningitis or meningoencephalitis.
* History of malignant neoplasms within 3 years prior to study screening or where there is current evidence of recurrent or metastatic disease.
* History of persistent cognitive deficits immediately following head trauma.
* History of inflammatory neurology disorders.
* History of autoimmune disease with potential for CNS involvement.
* MRI scan at screening showing a single area of cerebral vasogenic edema, superficial siderosis, or evidence of a prior macrohemorrhage, or showing more than four cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite").
* MRI examination cannot be done for any reason, including metal implants contraindicated for MRI studies and/or severe claustrophobia.
* Significant hearing or visual impairment or other issues judged relevant by the investigator preventing to comply with the protocol and to perform the outcome measures.
* Severe infections or a major surgical operation within 3 months prior to screening.
* History of chronic or recurrent infections judged to be clinically significant by the investigator.
* History or presence of immunological or inflammatory conditions which are judged to be clinically significant by the investigator.
* Celiac disease not on a gluten free diet for at least 3 months prior to study screening.
* Chronic benign skin pathologies, unless viewed as clinically insignificant in the investigator's opinion.
* Any vaccine received within the past 2 months before baseline, except influenza vaccine which if indicated must be given at least 2 weeks prior to baseline.
* Clinically significant arrhythmias or other abnormalities on ECG at screening. (Minor abnormalities documented as clinically insignificant by the investigator will be allowed.)
* Clinically significant abnormal vital signs including sustained sitting blood pressure greater than 160/90 mmHg.
* In the opinion of the site investigator, deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, that are judged to be clinically significant.
* Subjects with treated hypothyroidism not on a stable dose of medication for at least 3 months prior to screening and having clinically significant abnormal serum T-4 and TSH at screening.
* Subjects with diabetes mellitus with an HbA1c of ≥ 8.0%.
* Subjects who have been receiving any experimental drug for Down Syndrome with a washout less than 30 days or less than five halflives of the drug, whichever is longer.
* Female subjects being pregnant as confirmed by serum testing at screening or planning to be pregnant or lactating.
* Female subjects not using a reliable method of contraception (unless abstaining).
* Patient receiving any anticoagulant drug, or aspirin at doses greater than 100 mg daily in the 7 days prior to lumbar puncture (in order to avoid risk of bleeding during scheduled or unscheduled lumbar puncture)
* Use of antidepressants other than SSRI/SNRIs at stable dose, antipsychotics (typical or atypical), GABA agonists (e.g. gabapentin), or stimulants (e.g. methylphenidate, modafinil). In exceptional cases, low doses of atypical antipsychotics (e.g. risperidone up to 0.5 mg/day or quetiapine up to 50 mg/day) or benzodiazepines are only allowed after review by the site principal investigator, in consultation with the project director and/or medical monitors.
* Current use of immunosuppressant or immunomodulating drugs or their use within the past 6 months prior to study screening. Current use of steroids or their use within the past 3 months prior to study screening.
* Use of Cholinesterase Inhibitor or use of Glutamatergic drugs (Topiramate, Memantine, Lamotrigine) if not on stable dose for at least 3 months prior to screening.
* Subjects who have donated blood or blood products during the 30 days prior to screening who plan to donate blood while participating in the study or within four weeks after completion of the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Rafii, MD, PhD, Study Director — USC Keck School of Medicine of the University of Southern California, San Diego
Locations (4):
- United States (4):
  - St. Joseph's Hospital and Medical Center - Barrow Neurology Clinics, Phoenix, Arizona
  - UCSD Adult Down Syndrome Program, La Jolla, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Access to de-identified, individual and trial -level data (analysis datasets), and other information (e.g., protocols) will be provided.
Supporting Information: Study Protocol, SAP
Access Criteria: These clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research and will be provided after review and approval of their research proposal, their Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). Data sharing shall be in accordance with ADCS' data sharing plan in its grant application and applicable NIH policy in effect at the time of the NIH award.
URL: https://www.adcs.org/

REFERENCES:
- [Derived] Rafii MS, Sol O, Mobley WC, Delpretti S, Skotko BG, Burke AD, Sabbagh MN, Yuan SH, Rissman RA, Pulsifer M, Evans C, Evans AC, Beth G, Fournier N, Gray JA, Dos Santos AM, Hliva V, Vukicevic M, Kosco-Vilbois M, Streffer J, Pfeifer A, Feldman HH. Safety, Tolerability, and Immunogenicity of the ACI-24 Vaccine in Adults With Down Syndrome: A Phase 1b Randomized Clinical Trial. JAMA Neurol. 2022 Jun 1;79(6):565-574. doi: 10.1001/jamaneurol.2022.0983. PMID 35532913

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty subjects were screened (signed the informed consent) but four participants were considered screen failures
Groups:
- ACI-24 300µg: Cohort 1: Low dose
- ACI-24 1000µg: Cohort 2: High dose
- Placebo: Placebo cohort 1 + cohort 2
Period: Overall Study
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Started | 6 | 6 | 4
Completed | 6 | 4 | 4
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The data of the 20 subjects who have signed the informed consent (ie including the screen failure subject) have been considered.
Groups:
- Screen Failure: Screen failure cohort 1 + cohort 2
- Total: Total of all reporting groups
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo | Screen Failure | Total
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (4.6) | 31.5 (4.9) | 33.0 (4.2) | 34.0 (2.6) | 32.9 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 2 | 11
  Male | 4 | 2 | 1 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 4 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 4 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 4 | 4 | 20
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.0 (9.9) | 39.9 (9.4) | 43.1 (12.7) | 42.8 (11.6) | 40.2 (10.1)
KBIT 2: IQ Composite [Mean (Standard Deviation); unit: IQ score] — The 20 subjects who have signed the informed consent (ie including the 4 screen failure subjects) have completed the KBIT 2.
  The KBIT 2 range score is from 40 to 160, lower score means a worse outcome
  IQ score | 44.2 (5.5) | 49.2 (9.5) | 46.0 (8.0) | 52.8 (18.9) | 47.8 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titer (Serum Anti-Aβ1-42 Free IgG) - Mean Absolute Value
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  The measure is expressed in Arbitrary Units per mL (AU/mL). AU/mL in a sample is obtained by back-calculation towards the standard curve.
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: Modified Intent to Treat Population (mITT)
Measure: Mean (Standard Deviation); unit: AU/mL (AU: Arbitrary Unit)
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
AU/mL (AU: Arbitrary Unit)
  Week 0 | 632.3 (570.9) | 335.4 (157.4) | 162.8 (84.5)
  Week 50 | 751.5 (825.6) | 434.3 (224.3) | 153.3 (140.7)

2. Secondary Outcome: Amyloid Beta 1-40 in Blood - Mean Absolute Value
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
ng/L
  Week 0 | 81.7 (56.6) | 138.5 (41.1) | 169.5 (43.5)
  Week 50 | 183.8 (18.7) | 186.2 (37.8) | 181.3 (11.2)

3. Secondary Outcome: CANTAB - MOT Latency Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Cambridge Neuropsychological Test Automated Battery (CANTAB), Motor Screening Task (MOT) is a cognitive scale to be completed by the subject.
  Range score from 0 to ∞, lower score means a better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  week 0 | 1784.5 (904.4) | 997.1 (271.8) | 1024.3 (193.9)
  Week 50 | 1781.2 (960.4) | 1046.3 (152.1) | 1002.1 (138.5)

4. Secondary Outcome: CANTAB - PAL First Attempt Memory Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Cambridge Neuropsychological Test Automated Battery (CANTAB), Paired Associate Learning (PAL) is a cognitive scale to be completed by the subject.
  Range score from 0 to 20, higher score means a better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  week 0 | 8.0 (5.1) | 9.2 (5.1) | 7.8 (5.3)
  Week 50 | 7.5 (4.1) | 6.7 (4.3) | 9.8 (4.6)

5. Secondary Outcome: Brief Praxis Test (BPT) - Total Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Brief Praxis Test (BPT) is a cognitive scale to be completed by the subject.
  Range score from 0 to 80, higher score means better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  Week 0 | 72.0 (5.8) | 73.7 (3.2) | 73.8 (5.6)
  Week 50 | 75.5 (4.8) | 77.5 (2.5) | 76.5 (2.5)

6. Secondary Outcome: Vineland II - Communication Domain Standard Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Vineland II is a behavioral questionnaire to be completed by the study partner of the subject.
  Range score from 0 to 113, higher score means a better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  Week 0 | 47.7 (10.2) | 59.3 (8.5) | 59.0 (5.3)
  Week 50 | 52.2 (11.3) | 65.2 (9.4) | 61.0 (6.8)

7. Secondary Outcome: Vineland II - Daily Living Skill - Domain Standard Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Vineland II is a behavioral questionnaire to be completed by the study partner of the subject.
  Range score from 0 to 114, higher score means a better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  Week 0 | 54.2 (9.9) | 68.3 (4.1) | 58.0 (9.3)
  Week 50 | 55.8 (11.4) | 72.8 (4.1) | 61.5 (13.5)

8. Secondary Outcome: Vineland II - Socialisation - Domain Standard Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Vineland II is a behavioral questionnaire to be completed by the study partner of the subject.
  Range score from 0 to 115, higher score means a better outcome
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  Week 0 | 64.3 (17.2) | 77.0 (9.1) | 59.0 (15.1)
  Week 50 | 66.7 (16.1) | 83.0 (10.4) | 70.3 (9.7)

9. Secondary Outcome: NPI - Total Score
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Neuropsychiatric Inventory (NPI) is a behavioral questionnaire to be completed by the study partner of the subject.
  Range score from 0 to 144, higher score means a worse outcome
Time Frame: Values at baseline (week 0) and week 50 are reported.
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale
  Week 0 | 4.5 (3.6) | 0.3 (0.8) | 8.5 (10.0)
  Week 50 | 1.5 (2.5) | 0.3 (0.8) | 4.0 (8.0)

10. Secondary Outcome: Clinical Global Impression of Change (CGIC) - Change From Baseline at Week 50
Description: All subjects who received at least 1 dose of the study treatment of either ACI-24 300 μg, ACI-24 1000 μg or placebo are considered.
  Clinical Global Impression of Change (CGIC) is a global assessment to be completed by the investigator.
Time Frame: Values at baseline (week 0) and week 50 are reported
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants
  Marked improvement | 0 | 0 | 1
  Moderate improvement | 1 | 0 | 1
  no change | 5 | 6 | 2

ADVERSE EVENTS:
Time Frame: The collection of Treatment Emergent Adverse Events (TEAEs) for an individual subject started after the first dose at baseline (Week 0) and finished at the end of the designated follow-up period at Week 96.
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Placebo Cohort 1: Cohort 1: Placebo
- Placebo Cohort 2: Cohort 2: Placebo
Arm/Group | ACI-24 300µg | ACI-24 1000µg | Placebo Cohort 1 | Placebo Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACI-24 300µg (N=6) | ACI-24 1000µg (N=6) | Placebo Cohort 1 (N=2) | Placebo Cohort 2 (N=2)
Infections and infestations (Infections and infestations) | 5 (18) | 3 (14) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 3 (5) | 3 (6) | 0 (0) | 1 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (5) | 1 (3) | 0 (0) | 2 (3)
General disorders and administration site conditions (General disorders) | 2 (2) | 2 (9) | 1 (1) | 1 (1)
Investigations (Investigations) | 2 (2) | 2 (3) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (5) | 3 (7) | 1 (1) | 0 (0)
Eye disorders (Eye disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vascular disorders (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study included a limited number of subjects, and, as a consequence, was not powered on cognition and clinical efficacy outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may freely publish and disseminate the results of the Study. However Institution shall only make a Publication once the Study has been completed. Institution shall send Sponsor any Publication 60 days prior to submission and Sponsor may make editorial changes to the Publication. Institution shall delete information that Sponsor considers as Confidential and Institution shall delay Publication for an additional 60 days to protect the potential patentability of an invention.

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT02738450/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT02738450/SAP_001.pdf